CLINICAL TRIAL: NCT06251986
Title: A Cross-sectional Study to Assess the Effectiveness and Safety of Ofatumumab (Kesimpta®) in Patients With Relapsing Multiple Sclerosis in the Spanish Clinical Practice: the CRONOS-MS Study.
Brief Title: A Cross-sectional Study to Assess the Effectiveness and Safety of Ofatumumab (Kesimpta®) in Patients With Relapsing Multiple Sclerosis in the Spanish Clinical Practice
Acronym: CRONOS-MS
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GES01
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: RMS; NIS; Spain; ofatumumab
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- ofatumumab: Subcutaneous ofatumumab in a real-world setting
  Interventions: Other: ofatumumab

INTERVENTIONS:
Other: ofatumumab — This is an observational study, there was no treatment allocation.

SUMMARY:
This was a non-interventional, cross-sectional, multicentric, and nationwide study, based on primary and secondary data collection.

DETAILED DESCRIPTION:
The present study aimed to characterize the use of subcutaneous ofatumumab in a real-world setting. Specifically, the investigation assessed the effectiveness, safety, and treatment adherence associated with subcutaneous ofatumumab in individuals with relapsing forms of multiple sclerosis (RMS) within the Spanish healthcare system.

The study used primary and secondary data collection. Primary data collection included information collected using PRO, clinical-reported outcomes (ClinRO), scales or tests and the interview during the study visit. Secondary data collection included existing data from electronic medical records (EMR) or paper-based medical records, collected as part of the routine follow-up of patients with RMS in the clinical practice.

Baseline was defined as the date of ofatumumab initiation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years.
2. Written informed consent.
3. Diagnosis of RMS per McDonald Criteria (2017).
4. Ofatumumab treatment in line with the European Kesimpta® summary of product characteristics (SmPC; i.e. adult patients with RMS with active disease defined by clinical or imaging features) during at least 12 months and patients who discontinued ofatumumab after receiving at least one dose with a minimum monitoring of 12 months.

Exclusion Criteria:

1. Currently participating in a clinical trial.
2. Not able/unlikely to complete with all study activities according to investigator's criteria.
3. Have a contraindication for ofatumumab use, according to the SmPC.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with relapsing forms of multiple sclerosis (RMS) with active disease
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Reductions in the Annualized relapse rate (ARR) | 12 months preceding the initiation of ofatumumab, Baseline
  ARR, defined as the total number of confirmed relapses that occurred during the observation period divided by the total number of patient-years, with the result standardized to a 1-year period.
  A relapse is defined as new or recurrent symptoms and objective typical findings of MS with a duration of at least 24 h, in the absence of fever or infection and preceded by a stable or improving neurological state for ≥ 30 days

SECONDARY OUTCOMES:
Reductions in the ARR in naïve vs previously treated patients | 12 months preceding the initiation of ofatumumab, Baseline
  ARR, defined as the total number of confirmed relapses that occurred during the observation period divided by the total number of patient-years, with the result standardized to a 1-year period.
  A relapse is defined as new or recurrent symptoms and objective typical findings of MS with a duration of at least 24 h, in the absence of fever or infection and preceded by a stable or improving neurological state for ≥ 30 days
Reductions in the ARR in previously treated with high-efficacy Disease-modifying treatments (DMT) vs previously treated with moderate-efficacy DMT | 12 months preceding the initiation of ofatumumab, Baseline
  ARR, defined as the total number of confirmed relapses that occurred during the observation period divided by the total number of patient-years, with the result standardized to a 1-year period.
  A relapse is defined as new or recurrent symptoms and objective typical findings of MS with a duration of at least 24 h, in the absence of fever or infection and preceded by a stable or improving neurological state for ≥ 30 days
Number of days from ofatumumab treatment initiation to first relapse | 12 months
  A relapse is defined as new or recurrent symptoms and objective typical findings of MS with a duration of at least 24 h, in the absence of fever or infection and preceded by a stable or improving neurological state for ≥ 30 days
Proportion of relapse-free patients | 12 months
  A relapse is defined as new or recurrent symptoms and objective typical findings of MS with a duration of at least 24 h, in the absence of fever or infection and preceded by a stable or improving neurological state for ≥ 30 days
Change in EDSS score | Baseline, month 6, month 12
  The Expanded Disability Status Scale (EDSS) is the most widely disability scale used in MS. The scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist.
Number of participants with radiological disease activity on the cranial MRI | Baseline, month 6, month 12
  Number of participants with presence of radiological disease activity on the cranial MRI
Percentage of participants reporting injection site reactions (ISR) | Baseline, month 6, month 12
  Percentage of participants reporting injection site reactions (ISR)
Percentage of patients with AEs leading to temporal or permanent discontinuation | Up to 12 months
  Percentage of patients with AEs leading to temporal or permanent discontinuation
Number of pregnancies and pregnancy outcome | Up to 12 months
  Number of pregnancies and pregnancy outcome
Proportion of participants with non-adherence | Up to 12 months
  Non-adherence, defined as skipping at least one dose during initial dosing (i.e. missing one weekly injections, defined as not receiving the dose within the established 7 and 14 days after the prior dose) or during maintenance dosing (missing one monthly injection, defined as not receiving the dose within the established month after the prior dose) as per SmPC.
Proportion of patients who discontinue ofatumumab during the observation period | Up to 12 months
  Proportion of patients who discontinue ofatumumab during the observation period
Scores on the Work Productivity and Activity Impairment (WPAI) questionnaire | Baseline
  The WPAI is an instrument to assess impairments in both paid work and unpaid work. Using six questions, it measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days.
  The first question is neutral. In the 2nd 3rd 5th and 6th questions a higher score means worse outcome. In the 4th question a higher score means better outcome.
Scores on the SDMT | Baseline
  Symbol Digit Modalities Test (SDMT) is a measure of sustained attention, processing speed, visual scanning, and motor speed. This test involves a coding schema consisting of nine abstract symbols, each paired with a number ranging from 1 to 9. The subject is required to scan the key and write down the number corresponding to each symbol as fast as possible. The score is the number of correctly coded items from 0-110 where higher scores indicate better result.
Scores on the Modified Fatigue Impact Scale-5 (MFIS-5) | Baseline
  The MFIS-5 measures the impact of fatigue on cognitive, physical, and psychosocial function. The MFIS-5 is a self-administered questionnaire with a 5-point Likert scoring system that best indicates how often fatigue has affected patients during the past 4 weeks: 'never', 'rarely', 'sometimes', 'often' and 'almost always', each scored 0-4, respectively. It consists of 5 of the 21 items of MFIS that most strongly correlate with the total MFIS score. The sum provides a total score from 0 to 20. Higher scores indicate a higher perception of fatigue.
Scores on the EuroQol-5 dimension (EQ-5D)-5L | Baseline
  The EQ-5D-5L is a generic measure for Health-related quality of life. It consists of two pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has five levels( 1=no problems to 5= extreme problems). A summary index with a maximum score of 1 can be derived from these five dimensions by conversion with a table of scores. The maximum score of 1 indicates the best health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. In the VAS, 100 indicates the best health status.
Scores on the Patients' Global Impression of Change (PGIC) scale completed by patients | Baseline
  The PGIC is a single, self-administered question asking respondents to rate how their condition has changed since a certain point in time. The PGIC will ask: "Since beginning treatment, how would you describe the change (if any) in activity limitations, symptoms, emotions and overall quality of life, related to your MS? Responses will range from 1= very much improved to 7= very much worse.
Scores on the Clinical Global Impressions (CGI) scale completed by physicians | Baseline
  The CGI provides an overall clinician-determined summary measure that considers all available information, including the patient's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the patient's ability to function.
  The CGI-Improvement will be used in this study. The clinician compares the patient's overall clinical condition to the one week period just prior to the initiation of medication use. The following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.
Scores on the Treatment Satisfaction Questionnaire for Medication (TSQM-9) | Baseline
  The TSQM-9 is a widely used generic measure to assess treatment satisfaction with their medication.
  The TSQM-9 uses nine of the 14 TSQM Version 1.4 items not including five TSQM questions related to side effects. The TSQM-9 encompasses three subscales that assess the patient's perception of medication effectiveness, convenience, and global satisfaction. Each TSQM-9 subscale consists of three items, with responses measured on a Likert scale ranging from 1 (low) to 7 (high). Subscale scores are usually transformed to a range from 0 to 100, with higher scores indicating greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Spain (25):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Palma, Balearic Islands
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Albacete, Castille-La Mancha
  - Novartis Investigative Site, Salt, Girona
  - Novartis Investigative Site, Logroño, La Rioja
  - Novartis Investigative Site, Fuenlabrada, Madrid
  - Novartis Investigative Site, Majadahonda, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Santa Cruz, Santa Cruz de Tenerife
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Alicante
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Burgos
  - Novartis Investigative Site, Cáceres
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Granada
  - Novartis Investigative Site, León
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18396